CLINICAL TRIAL: NCT00712400
Title: Effects of Latanoprost on Choroidal Blood Flow Regulation in Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: OPHT-070703
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Ocular Physiology; Intraocular Pressure; Regional Blood Flow
Keywords: Latanoprost; Choroidal Blood Flow; Intraocular Pressure
MeSH Terms: interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Latanoprost 0.005%, Xalatan®
  Interventions: Drug: Latanoprost 0.005%, Xalatan®
- 2 (Placebo Comparator): Vehicle to latanoprost (eyedrops containing the same stabilizers as latanoprost, but no active drug)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Latanoprost 0.005%, Xalatan® — Substance: Latanoprost 0.005%, Xalatan® (Pharmacia Austria Ges.m.b.H. Oberlaaer Straße 251, 1101 Vienna) Dosage form: topical application in one eye Dosage: 1 drop in the evening for 14 days
  Arms: 1
Drug: Placebo — Substance: Vehicle to latanoprost (eyedrops containing the same stabilizers as latanoprost, but no active drug) Dosage form: topical application in one eye Dosage: 1 drop in the evening for 14 days
  Arms: 2

SUMMARY:
Latanoprost is a synthetic prodrug of 17-phenyl-substituted prostaglandin F2α analog. Used at a dose of one drop per day, it has been reported to produce a 30 to 35% reduction in intraocular pressure. Its mechanism of activation involves augmentation of the eye's natural uveoscleral outflow capacity .

There is evidence that ocular blood flow plays a role in the clinical course of glaucoma. Glaucoma medication that lowers IOP simultaneously increases ocular blood perfusion pressure, which in turn may increase ocular blood flow.

This could well contribute to the partially contradicting results concerning ocular hemodynamic effects of latanoprost. In vitro studies indicate that latanoprost has no effect on ocular vascular tone in therapeutical doses. By contrast, it has been reported in several studies that latanoprost 0.005% increases pulsatile ocular blood flow in patients with primary open angle glaucoma and normal tension glaucoma. This increase in pulsatile ocular blood flow mainly reflects an increase in the choroidal circulation.

Little is known about the potential effect of latanoprost on choroidal blood flow regulation in humans. The present study therefore tries to elucidate whether treatment with latanoprost may alter choroidal blood flow regulation during artificial changes in ocular perfusion pressure. In addition, the present study aims to clarify whether the change in choroidal blood flow after latanoprost administration are due to direct vasoactive effects or due to the increase in ocular perfusion pressure. The second alternative may have important implications on our understanding of glaucoma treatment, because reduction of IOP may then per se result in normalization of ocular blood flow regulation.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Ametropia >= 3 dpt
* Iris bicolor

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-06; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Choroidal pressure-flow relationship | in total 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Derived] Boltz A, Schmidl D, Weigert G, Lasta M, Pemp B, Resch H, Garhofer G, Fuchsjager-Mayrl G, Schmetterer L. Effect of latanoprost on choroidal blood flow regulation in healthy subjects. Invest Ophthalmol Vis Sci. 2011 Jun 22;52(7):4410-5. doi: 10.1167/iovs.11-7263. PMID 21498617